CLINICAL TRIAL: NCT02060409
Title: Prognostic Molecular Markers Determined by Using Gene Expression Profiling in Patients With Myelodysplastic Syndrome
Brief Title: Prognostic Molecular Markers in Patients With Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jun Ho Jang, Jun Ho Jang, Samsung Medical Center
Other Study IDs: 2012-01-081-003
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; decitabine; spliceosome mutation
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Genomic DNA extracted from bone marrow aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- spliceosome: patient who have available data for spliceosome mutation status
  Interventions: Genetic: spliceosome

INTERVENTIONS:
Genetic: spliceosome — spliceosome mutations

SUMMARY:
In the era of hypomethylating agent in MDS treatment, the investigators aimed to investigate the prognostic impact of mutations in spliceosome machinery genes (SRSF2, U2AF1, and ZRSR2) on the outcomes of 1st line decitabine treatment in MDS.

DETAILED DESCRIPTION:
A number of studies have tried to investigate clinical impact of mutations in spliceosomal machinery genes in MDS but they failed to demonstrate a consistent prognostic relevance. Moreover, the clinical impact of these mutations on the outcomes of hypomethylating agent treatment in MDS has never been explored yet. The investigators investigated the prognostic impact of mutations in spliceosome machinery genes (SRSF2, U2AF1, and ZRSR2) on the outcomes of 1st line decitabine treatment in MDS.

ELIGIBILITY:
Inclusion Criteria:

* de novo MDS patients were included in the study who had received 1st line decitabine treatment and had adequate genomic DNA from pretreated bone marrow samples

Exclusion Criteria:

* therapy-related MDS

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: de novo MDS patients were included in the study who had received 1st line decitabine treatment and had adequate genomic DNA from pretreated bone marrow samples
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
overall survival | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Jang, MD PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hong JY, Seo JY, Kim SH, Jung HA, Park S, Kim K, Jung CW, Kim JS, Park JS, Kim HJ, Jang JH. Mutations in the Spliceosomal Machinery Genes SRSF2, U2AF1, and ZRSR2 and Response to Decitabine in Myelodysplastic Syndrome. Anticancer Res. 2015 May;35(5):3081-9. PMID 25964599